CLINICAL TRIAL: NCT01424046
Title: Evaluation of Differing Type 1 Diabetes Regimens in Youth in the Developing World
Brief Title: Health Care for Type 1 Diabetes in Developing World
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National University, Rwanda (Other); Association Rwandaise des Diabetiques (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC4 pitt 1; RC4DK090809 (NIH)
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; basal insulin; developing world; comparative effectiveness
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- basal insulin approach (Experimental): Participants will be treated primarily with a daily basal insulin injection ( glargine) with later introduction of prandial coverage with a shortacting insulin.
  Interventions: Drug: basal insulin glargine
- standard therapy (Active Comparator): Participants will continue current mixed insulin management and education
  Interventions: Drug: standard therapy

INTERVENTIONS:
Drug: basal insulin glargine — Individuals assigned to this arm will initially receive a basal insulin injection daily and gradually be introduced to meal time coverage of blood sugar with additional short acting insulin. Education will like wise proceed in a stepwise manner.
  Other Names: Lantus
  Arms: basal insulin approach
Drug: standard therapy — Participants will continue with current mixed insulin treatment using NPH , or lente, and regular insulin .
  Arms: standard therapy

SUMMARY:
This study is a pilot 2-armed, randomized, open label, clinical trial evaluating the effectiveness of a basal approach to diabetes management as compared to the current standard treatment (regular/NPH).

Patients seen at the Association Rwandaise des Diabetiques (ARD) will be invited to participate in the study and consent will be obtained by the investigation team. This will continue until 40 patients have been enrolled at which time recruitment will be started at a provincial hospital, at which 10 further participants will be recruited. Participants will be consenting to 1) Randomization to basal or current insulin treatment arm and 2) Permission for use of clinical data for research.Participants will be followed every six months for a period of 24 months. The first 6 months will be a wash in period and participants will be randomised (1/1) to their treatments at the 6 month visit.

DETAILED DESCRIPTION:
All participants will be provided with the consent form (that has been translated into the native language of Kinyarwandan) by the investigators and consent will be obtained from the participant if they are aged 18 and older or by parents/guardians if they are under 18 years. For those aged 14 - 17 years a child assent will be obtained. For those who are unable to read the consent form a patient advocate who will read this form to them and answer any questions a potential participant may have. Each person will have time and space to review all of the study information and they will be informed that participation is completely voluntary and that they will continue to receive their normal care if they do not wish to participate. At this visit the following data will be extracted from their clinical files by a research assistant under the supervision of Prof Kakoma:

At all 6 monthly visits (V1-V4), data from the participants' regular clinical visits (based on the annual evaluation form for the Life For a Child program) will be extracted. This includes HbA1c and microalbuminuria data collection, as well as documentation of: insulin regimen, incidents of severe hypo- and hyper-glycemia, symptoms of hyperglycemia, current schooling level, number of school days missed due to diabetes, self-rating of diabetes control, height, weight, blood pressure, and a basic neurological examination (vibratory sensation of great toe and monofilament testing). Information will be abstracted by research assistants from the National University of Rwanda (NUR), and education and management functions will be carried out by nurses from the ARD that will be trained by Drs Orchard and Edidin.

Each enrolled participant will be followed for a six month period post enrollment on their current treatment regimen so the impact of being enrolled in a study rather than an effect of their treatment, can be assessed.

All participants will be supplied with a glucose meter and sufficient strips to test daily. These results will also be made available to and reviewed by the ARD staff and will be used for further dose adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes being treated by the Association Rwandese des Diabetiques
* Resident of Rwanda

Exclusion Criteria:

* life expectancy less than three years
* requiring additional diabetes therapy beyond the scope of the trial

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | one year
  The primary outcome is the level of blood sugar control after 1 years treatment as determined by the Hb A1c test

SECONDARY OUTCOMES:
Microalbuminuria | one year
  Microalbuminuria, the leakage of abnormal amounts of protein in the urine is a major complication of type 1 diabetes and the prevalence of this in the two groups is a secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Trevor J Orchard, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Association Rwandese des Diabetiques, Kigali, Kigali Provence, Rwanda